CLINICAL TRIAL: NCT06606964
Title: The Influence of the Lower Limb Components on Genu Varum in Football Players: a Full Leg Length Magnetic Resonance Imaging Study
Brief Title: The Influence of the Lower Limb Components on Genu Varum in Football Players
Status: Completed | Type: Observational
Sponsor: Tuba Melekoğlu (Other)
Responsible Party: Sponsor-Investigator, Tuba Melekoğlu, Assoc. Prof., Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: KAEK-917
Record Dates: First submitted 2024-09-16; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Genu Varum; Football Players
Keywords: Genu varum; Knee joint; Mechanical axis deviation; Isokinetic strength; Football players
MeSH Terms: conditions — Genu Varum | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Football players with genu varum: Football players with genu varum leg alignment
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Other: Isokinetic Strength
- Football players without genu varum: Football players with normal lower extremity alignment
  Interventions: Diagnostic Test: Magnetic Resonance Imaging; Other: Isokinetic Strength

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — The MRI examinations were conducted using a 1.5 Tesla closed MRI system with a body coil and spine coil. The participants' knees were positioned in full extension and their feet were in a neutral position during imaging. The scan was performed from the anterior superior iliac spine to the tip of the toes, and both legs were included in the field of view
Other: Isokinetic Strength — The strength of the concentric knee extensor-flexor and concentric hip abductor-adductor muscles was measured using an isokinetic dynamometer at two different angular velocities: 60˚/sec and 180˚/sec. Three repetitions were performed at 60˚/sec, and five repetitions were performed at 180˚/sec. To calculate the H/Q ratio, we divided the peak concentric torque of the hamstrings by that of the quadriceps during the same contraction velocity. Similarly, to determine the Add/Abd ratio, we divided the peak concentric torque of the adductors by that of the abductors during the same contraction velocity

SUMMARY:
Objectives: To evaluate lower extremity alignments in football players with and without genu varum using magnetic resonance imaging (MRI), to determine the mechanisms underlying malalignment and the factors contributing to it.

Methods: This is a prospective case-control study with football players with/without lower extremity malalignment. Full-length lower extremity MRI was used to evaluate the lower extremity alignment parameters. In addition, the isokinetic strength of the concentric knee extensor-flexor and concentric hip abductor-adductor muscles was measured using an isokinetic dynamometer at two different angular velocities: 60˚/sec and 180˚/sec. The investigators created a logistic regression model to investigate whether the alignment parameters used to evaluate lower extremity alignment in football players are risk factors for the development of genu varum.

DETAILED DESCRIPTION:
Genu varum deformity is a common condition among football players, occurring in 73% of cases . Previous studies have shown that football players are at a higher risk of developing genu varum than athletes in other sports . Genu varum can have a negative impact on an athlete&#39;s physical abilities by disrupting static and dynamic balance through alterations in the gravitational axis of the lower extremities. In addition, genu varum can damage the tibiofemoral articular cartilage, increasing the risk of knee osteoarthritis later in life . It is also associated with several intra-articular pathologies, including meniscal lesions, anterior knee pain, and anterior cruciate ligament injuries . Therefore, it is important to understand the cause of this deformity and take protective-corrective measures for football players.

In recent years, researchers have studied the relationship between genu varum and football participation. Researchers have used various methods, including the caliper, goniometer, and photographic technique, to analyze deformities. However, these methods have limitations, making it difficult to examine etiological factors and differences in anthropometric components . In a study conducted by Colyn, Arnout, Verhaar and Bellemans 6, a comparison was made between football players and other athletes and non-athletes using digital radiology measurements. The findings indicated that male football players exhibited genu varum, with the proximal tibia identified as the primary factor determining this. Similarly, Krajnc and Drobnič studied lower limb alignment in asymptomatic adult professional football players and found that the proximal tibia was the source of varus deformity. However, it has been suggested that additional research is required to fully comprehend the involved mechanisms. Furthermore, Witvrouw, Danneels, Thijs, Cambier and Bellemans 9proposed that an imbalanced strength distribution between the adductor and abductor muscles may result in genu varum in football players. This is because kicking, a frequent activity in football, often strengthens the adductor muscles, which can alter the average adductor/abductor strength ratio. However, the authors note that no data on the adductor/abductor strength of football players is available in the literature. They suggest further research to address this knowledge gap.

Asymmetrical movements in football, resulting from the difference between the kicking and supporting legs, may lead to different mechanisms causing genu varum formation in the dominant and non-dominant legs. It is crucial to acknowledge that not all football players exhibit varus knee alignment. Consequently, in order to ascertain the mechanisms that contribute to the formation of genu varum, it is essential to conduct a comparative analysis between football players exhibiting and those lacking a varus deformity. This comparison can assist in identifying the mechanisms that cause genu varum in football players and the factors likely to contribute to these mechanisms. The study had three objectives: (i) to evaluate lower extremity alignments in football players with and without genu varum using magnetic resonance imaging (MRI), (ii) to determine the mechanisms underlying malalignment and the factors contributing to it; and (iii) to investigate the relationship between lower extremity alignment and isokinetic strength.

ELIGIBILITY:
Inclusion Criteria:

* Healthy football players who currently play for a professional football club
* Aged 16-19
* Have at least five years of football experience
* Train five days a week
* Participating in official matches.

Exclusion Criteria:

* History of musculoskeletal disease
* History of postural disorders
* History of previous surgery for lower extremity sports injuries
* History of fractures of the long bones of the lower extremity

Ages: 16 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study participants were selected from otherwise healthy football players aged 16-19 who currently play for a professional football club, have at least five years of football experience, train five days a week, and participate in official matches.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Mechanical axis deviation (MAD) | From enrollment to the end of measurements at 3 weeks
  The mechanical axis is a line connecting the center of the femoral head to the center of the ankle (center of the dome of the talus). A line was drawn from the center of the femoral head to the center of the ankle and the intersection of this line with the knee joint line was marked. The perpendicular distance from this intersection point to the center of the patella was measured as MAD.
Femoral anteversion (FA) | From enrollment to the end of measurements at 3 weeks
  On the axial images of the hip/pelvis covering the femoral head and neck, a line is drawn between the center of the femoral head and center of the femoral neck to calculate the uncorrected femoral anteversion angle. To correct for distal femoral rotation, another line is drawn along the posterior border of the femoral condyles to calculate the angle. Positive degrees between the femoral neck and the distal femoral axis are called femoral antetorsion; negative values were considered as femoral retrotorsion.
Medial proximal tibial angle (MPTA) | From enrollment to the end of measurements at 3 weeks
  The MPTA was defined as the medial angle between the proxsimal tibial joint line and the mechanical axis of the tibia. The proximal joint orientation line of tibia was drawn. A line was also drawn from the midpoint of the ankle to the midpoint of the knee on the tibial joint line. The angle between these two lines was measured.
Tibial torsion (TT) | From enrollment to the end of measurements at 3 weeks
  Proximal tibial axis (PTA) was placed along the posterior cortex of the tibial head at the level of condyls proximal to the fibular head. Distal tibial axis (DTA) was placed to the articular aspects of the medial and the lateral malleolus below the talar surface. The tibial torsion was calculated as the angle between the PTA and the DTA.
Tibial tubercle-trochlear groove (TT-TG) distance | From enrollment to the end of measurements at 3 weeks
  Firstly, transverse image that depicted a complete cartilaginous trochlea was used to determine the deepest point within the trochlear groove. A line was drawn through the deepest point of the trochlear groove, perpendicular to the posterior condylar tangent. Another line was drawn in parallel to the trochlear line through the most anterior portion of the tibial tubercle. Tibial tuberosity-trochlear groove distance was measured as the distance between these 2 lines.
Tibial tubercle-posterior cruciate ligament (TT-PCL) | From enrollment to the end of measurements at 3 weeks
  The TT-PCL distance was measured on axial images between the patellar tendon insertion midpoint and the medial border of the posterior cruciate ligament at its tibial insertion, parallel to the dorsal tibia condylar line.
Joint line convergence angle (JLCA) | From enrollment to the end of measurements at 3 weeks
  The mechanical axis line of femur was drawn, and then the knee joint line in the frontal plane was determined. The angle between these two lines was measured.
Hip-knee-ankle angle (HKA) | From enrollment to the end of measurements at 3 weeks
  The measurement was taken of the angle formed between the mechanical axis of the femur and tibia.
Mechanical lateral distal femoral angle (mLDFA) | From enrollment to the end of measurements at 3 weeks
  The distal joint orientation line of femur was drawn. A second line was drawn from the center of hip to the knee's midpoint at the femoral knee joint line (femoral mechanical axis). The angle between these two lines was measured.
Quadriceps femoris angle (Q angle) | From enrollment to the end of measurements at 3 weeks
  The angle between the lines connecting the anterior superior iliac spine (ASIS) to the midpoint of the patella, and from there to the tibial tubercle was measured.

SECONDARY OUTCOMES:
Isokinetic strength | From enrollment to the end of measurements at 3 weeks
  The strength of the concentric knee extensor-flexor and concentric hip abductor-adductor muscles was measured using an isokinetic dynamometer at two different angular velocities: 60˚/sec and 180˚/sec.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Melekoglu, Phd, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University Faculty of Sport Sciences, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during the current study will be available upon request from corresponder author Tuba Melekoğlu
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The datasets generated during the current study will be available upon request from publishing date
Access Criteria: The datasets generated during the current study will be available for researchers

REFERENCES:
- [Background] Asadi K, Mirbolook A, Heidarzadeh A, Mardani Kivi M, Emami Meybodi MK, Rouhi Rad M. Association of Soccer and Genu Varum in Adolescents. Trauma Mon. 2015 May;20(2):e17184. doi: 10.5812/traumamon.17184. Epub 2015 May 25. PMID 26290852
- [Derived] Isin A, Kose O, Ak E, Emir Yetim E, Cevikol C, Melekoglu T. The influence of the lower limb components on genu varum in football players: a full leg length magnetic resonance imaging study. BMC Sports Sci Med Rehabil. 2025 Feb 25;17(1):25. doi: 10.1186/s13102-025-01075-9. PMID 40001230